CLINICAL TRIAL: NCT00982241
Title: Prospective Intervention Study of Drink Advice in Overactive Bladder Syndrome (OAB)
Brief Title: Overactive Bladder (OAB) Drink Advice Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrolling participants
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OABdrinkstudy
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2009-09

CONDITIONS: Overactive Bladder Syndrome
Keywords: OAB; urine; osmolality; urge; fluid intake; PPIUS; urge score; bladder
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- normal fluid intake (Active Comparator): 1500 ml /day (+/- 300 ml) for 2,5 days
  Interventions: Dietary Supplement: water
- high fluid intake (Active Comparator): 2400 ml/day (+/- 300 ml )for 2,5 days
  Interventions: Dietary Supplement: water
- low fluid intake (Active Comparator): fluid intake 900 ml/day (+/- 300ml) for 2,5 days
  Interventions: Dietary Supplement: water

INTERVENTIONS:
Dietary Supplement: water — drinking water / normal dietary fluids for oral intake

SUMMARY:
The researchers want to investigate how fluid intake influences the symptoms of OAB. The researchers will recruit 45 patients with OAB and randomize them (blind) in 3 groups (low/normal/high fluid intake). Patients will follow this drink pattern for 2-5 days, while filling in an standard micturation diary for 2 days. This micturation diary is coupled to: collection of multiple urine samples, urine pH measurements, and a Perception of Intensity of Urgency Scale (PPIUS) scoring table. All this is collected by the patients themselves. Urine samples will be analysed for osmolality by the clinical chemistry department.

ELIGIBILITY:
Inclusion Criteria:

* OAB patients

Exclusion Criteria:

* benign prostatic hyperplasia
* neurogenic detrusor overactivity
* urine tract infection
* anticholinergics
* intravesical botulin toxin
* cardiac failure
* renal insufficiency
* sacral neurostimulation
* percutaneous neurostimulation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
urine osmolality | 2 days
PPIUS urge-score | 2 days

SECONDARY OUTCOMES:
urine pH | 2 days
PPIUS urge score | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: John Heesakkers, dr. MD, Study Chair — dept of Urology, Radboud University Nijmegen Medical Centre
Locations (1):
- Dept. of Urology, Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands